CLINICAL TRIAL: NCT02061878
Title: A Randomized Controlled Study to Evaluate the Effect of Bexarotene - an RXR Agonist - on Beta-Amyloid and Apolipoprotein E Metabolism in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Bexarotene on Beta-Amyloid and Apolipoprotein E Metabolism in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReXceptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: REXCEPTOR-101
Record Dates: First submitted 2014-02-05; First posted 2014-02-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer's Disease
Keywords: ApoE; beta-amyloid
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — Bexarotene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bexarotene (Experimental): The subjects will be administered three (3) capsules of Targretin™ (75 mg/capsule) on a twice daily basis (450 mg/day) for five days
  Interventions: Drug: Bexarotene
- Placebo (Placebo Comparator): The subjects will be administered three (3) capsules of Avicel PH on a twice daily basis (450 mg/day) for five days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bexarotene — Marketed product Targretin® soft gelatin capsule (75mg/capsule) is over-encapsulated in a size AA-el Swedish orange capsule. The subjects will be administered three (3) capsules of Targretin™ (75 mg/capsule) on a twice daily basis (450 mg/day) for five days.
  Other Names: Targretin®
  Arms: Bexarotene
Drug: Placebo — The subjects will be administered three (3) capsules of Avicel PH on a twice daily basis (450 mg/day) for five days.
  Other Names: Avicel PH
  Arms: Placebo

SUMMARY:
The primary objective of this proof of mechanism pilot clinical trial is to determine if the RXR agonist bexarotene acts in humans to alter the CSF levels of apoE and alter the clearance of Amyloid-Beta

DETAILED DESCRIPTION:
This is a double blinded, investigational drug study designed to measure the effect of bexarotene on the clearance of Aβ total and production of apoE in the human brain of young, healthy individuals with the APOE3/3 genotype. From the date of initial subject recruitment to the issuance of a final study report and closeout activities, the expected total study duration is 6 to 10 months.

Each participant will be screened for eligibility and randomized to receive either oral bexarotene or placebo control ("Test Article").The study has the potential to demonstrate the pharmacodynamic properties of a novel treatment approach to Alzheimer's disease. The primary biomarker measurements obtained from this study are believed to be highly dynamic and able to provide a rapid read-out of the biologic activity of the candidate therapeutic under study. In addition, exploratory analysis will involve a proteomics-based screen to identify proteins within both blood and CSF that are induced by the Test Article, thereby potentially identifying new biomarkers that can be used in future clinical trials to demonstrate bexarotene action and target engagement.

ELIGIBILITY:
Inclusion Criteria:

* Young healthy adults (age 21-50)
* APOE3/3 genotype

Exclusion Criteria:

* Contraindications for blood or CSF sampling
* Bleeding disorder or taking anticoagulants/antiplatelets
* Chronic active infection
* Blood donation within the past month
* Active drug/alcohol dependence or abuse history with in the last 12 months
* Thyroid dysfunction
* High triglycerides (>3.5 mmol/L)
* High cholesterol (>4.0 mmoL/L)
* Leukopenia, including low neutrophil count (<3 x 10^9/L)
* Neurological or psychiatric disorders
* Homeless or prisoner
* Pregnancy
* Incapable of self-informed consent
* Blood borne disease (HIV, Hepatitis)
* Actively smoking and incapable of using nicotine patches
* Known drug allergy to pain medication or local anesthetic
* Subjects that have participated in another study in the last 30 days
* Abnormalities in lumbar spine previously known within 12 months
* APOE2 or APOE4 allele
* Abnormal EKG

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area under the effect curve for newly generated beta-Amyloid (clearance phase), | 21 - 48 hr
  Area under the effect curve from 21-48h for newly generated beta-Amyloid (clearance phase), which is computed for each individual as the area under the curve of the clearance portion of the labeled beta-Amyloid curve between 21 hour and 48 hours, normalized by plasma free leucine levels.

SECONDARY OUTCOMES:
Fractional clearance rate of beta-Amyloid peptide in CNS | 21 - 36 hrs
  Fractional clearance rate (FCR) of beta-Amyloid peptide in CNS, computed for each individual as the slope of the natural logarithm of the clearance portion of the labeled beta-Amyloid curve between 21 hours and 36 hours 2) AUEC0-24 of apoE: Area under the effect curve from 0-24h for newly generated apoE (production phase) 3) Fractional synthesis rate (FSR) of apoE protein in CNS 4) Aβ and apoE concentrations: CSF beta-Amyloid and apoE concentrations for each time point 5)Size of apoE-containing high density lipoprotein particles in CSF as assessed by native PAGE 6) Labeled/Unlabeled Leu ratio (% of 13C6 Leu) in plasma and CSF for 48 hours following start of 13C6 Leu administration 7) Bexarotene concentrations in blood and CSF 8) Plasma beta-Amyloid total and apoE concentrations at baseline compared to final plasma beta-Amyloid total and apoE concentrations

OTHER OUTCOMES:
Exploratory Endpoint | 5 days
  AUEC0-18 for newly generated beta-Amyloid (production phase)

CONTACTS AND LOCATIONS:
Overall Officials: Craig T Curtis, MD, Principal Investigator — Compass Research
Locations (1):
- Compass Research, Orlando, Florida, United States

REFERENCES:
- [Derived] Ghosal K, Haag M, Verghese PB, West T, Veenstra T, Braunstein JB, Bateman RJ, Holtzman DM, Landreth GE. A randomized controlled study to evaluate the effect of bexarotene on amyloid-beta and apolipoprotein E metabolism in healthy subjects. Alzheimers Dement (N Y). 2016 Jun 17;2(2):110-120. doi: 10.1016/j.trci.2016.06.001. eCollection 2016 Jun. PMID 29067298